CLINICAL TRIAL: NCT00403884
Title: Selective RPE Laser Treatment (SRT) for Various Macular Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Dr. Werner Jackstaedt Foundation (Unknown)
Responsible Party: PD Dr. med. Carsten Framme, FEBO, MHM, University Eye Hospital Regensburg
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: University Eye Hospital SRT
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2006-11

CONDITIONS: Age-Related Macular Degeneration; Diabetic Maculopathy; Central Serous Chorioretinopathy
Keywords: Drusen; Geographic atrophy; diabetes; macular edema; laser; retinal pigment epithelium
MeSH Terms: conditions — Macular Degeneration; Central Serous Chorioretinopathy; Geographic Atrophy; Diabetes Mellitus; Macular Edema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Selective RPE laser treatment — interventional SRT laser treatment
  Other Names: SRT vario, Medical Laser Center, Luebeck, Germany

SUMMARY:
In this prospective clinical study SRT is performed with various pulse durations at 1.7µs and additionally 200ns to evaluate the different clinical effects of both laser regimens. The macular diseases to be treated are drusen maculopathy and geographic atrophy due to age-related macular degeneration as well as diabetic macular edema and central serous chorioretinopathy.

The beneficial effect in laser treatment is thought to be associated with the restoration of a new barrier of retinal pigment epithelium cells. If this theory is true, the destruction of the photoreceptors causing visual field defects would be only an unwanted and unnecessary side effect. Thus, SRT is able to avoid these unintentional side effects and to achieve the benefit by just treating the RPE.

In this study the clinical effect of SRT for these diseases is evaluated on a long-term basis.

DETAILED DESCRIPTION:
Conventional laser photocoagulation has been shown to be beneficial in a variety of retinal diseases like age related macular degeneration (AMD), diabetic maculopathy (DMP), diabetic retinopathy (DRP) or central serous retinopathy (CSR). There are several hints that the positive effect is mediated by the RPE. The RPE is the main target of laser energy due to its high amount of melanosomes and absorbs about 50 to 60 % of the energy applied to the retina. Today conventional retinal laser treatment is performed using the continuous-wave argon laser (514 nm). Generally the exposure times are longer than 50 ms, typically 100 to 200ms. After application of the laser energy onto the retina usually an ophthalmoscopically visible grayish-white lesion results from thermal heat conduction. Histologically a destruction of the RPE, which is the primary absorption site, occurs, leading to an irreversible destruction of the outer and inner segments of the neuroretina due to thermal denaturation.

The effect of laser treatment to the fundus was studied by several groups. In vivo it could be observed that argon laser photocoagulation of the monkey- and human fundus causes necrosis of the RPE and a detachment of the RPE from Bruch´s membrane, budding of individual RPE cells and a multilayered RPE formation in the area of laser irradiation by seven days after treatment. Histologic sections revealed that by irradiating the RPE with a conventional argon laser the whole area of the cells is destroyed and the choriocapillaris as well as the vessels of the choroid are damaged. After laser photocoagulation RPE cells migrate and proliferate to cover the defect. In vivo after mild coagulations as usually performed in macular coagulation the RPE barrier gets intact again.

Several macular diseases are thought to be caused only by a reduced function of the RPE cells. Therefore a method for the selective destruction of the RPE cells without causing adverse effects to choroid and neuroretina, especially to the photoreceptors, seems to be an appropriate treatment (SRT). The selective effect on RPE cells, which absorb about 50% of the incident light due to their high melanosome content has been demonstrated using 5 µs argon laser pulses at 514nm with a repetition rate of 500 Hz. By irradiating the fundus with a train of µs laser pulses it was possible to achieve high peak temperatures around the melanosomes. This led to a destruction of the RPE, but only a low sublethal temperature increase in adjacent tissue structures. This selective destruction of the RPE cells sparing the photoreceptors without causing laser scotoma has been proven by histologic examinations at different times after treatment. The first clinical trial using a Nd:YLF laser system with a pulse duration of 1,7µs (100 pulses, 100 and 500 Hz) also proved the concept of selective RPE destruction and demonstrated the clinical potential of this technique. However, one of the problems concerning selective RPE laser destruction is the inability to visualize the laser lesions. Therefore it is necessary to perform fluorescein angiography after treatment to confirm the laser success and to make sure that sufficient energy was used. Since dosimetry of such laser lesions is not known, test lesions with various energy and numbers of pulses in non-significant areas of the macula - usually at the lower vessel arcade - have to be applied to elucidate the energy levels required for treatment. If the RPE is damaged, or the tight junctions of the RPE barrier are broken, fluorescein from angiography can pool from the choriocapillaris into the subretinal space. Thus fluorescein angiography has been used to detect a break of the RPE barrier. However, fluorescein angiography is an invasive method and has as already described a potential risk for allergic reactions because of the intravenous injection of the fluorescein dye.

The damage mechanism in SRT is more a thermo-mechanical one than a purely thermal one as in conventional laser treatment due to the short-duration laser pulses in the microsecond-regime. Thus, microbubble formation around the melanosomes inside the RPE cell occurs during treatment, probably leading to disruption of the cell; this is in contrast to thermal denaturation in conventional laser photocoagulation. The formation of microbubbles around the strong absorbing melanosomes inside the RPE has been proofed as damage mechanism during irradiation of the RPE with µs laser pulses. If energy is absorbed and converted to heat the thermoelastic expansion of the absorbing medium will generate an opto-acoustic (OA) transient. During irradiation of RPE with µs laser pulses a classical thermoelastic transient will be emitted. Due to the formation and collapse of microbubbles around the melanosomes during a successful SRT treatment, additional OA bubble transients will be emitted. This is analogous to the emission of acoustic transients during formation and collapse of cavitation bubbles. An OA based on-line dosimetry system can differentiate between a pure thermoelastic transient in a subthreshold irradiation and OA bubble transients superimposed to the pure thermoelastic transients in case of a successful treatment irradiation. Thus, SRT can clinically be guided by this specific OA detection system.

In this prospective clinical study SRT is performed with various pulse durations at 1.7µs and additionally 200ns to evaluate the different clinical effects of both laser regimens, which were already determined to be safe in animal experiments. The macular diseases to be treated are drusen maculopathy and geographic atrophy due to age-related macular degeneration as well as diabetic macular edema and central serous chorioretinopathy.

The beneficial effect in laser treatment of diabetic macular edema is thought to be associated with the restoration of a new barrier of retinal pigment epithelium cells. A similar effect is postulated in the treatment of drusen, central serous retinopathy and macular edema after vein occlusion. If these latter theories are true, the destruction of the photoreceptors causing visual field defects would be only an unwanted and unnecessary side effect. Thus, SRT is able to avoid these unintentional side effects and to achieve the benefit by just treating the RPE.

In this study the clinical effect of SRT for these diseases is evaluated on a long-term basis. For diabetic macular edema previously non-treated eyes with focal or diffuse macular edema are randomized to SRT or conventional treatment. Best corrected visual acuity has to be at least 0.1 and no central ischemia must be present. The endpoint is visual acuity and reduction of edema as determined by fundus photography, angiography and optical coherence tomography. Regarding central serous chorioretinopathy visual acuity decay should last longer than 2 months with angiographically seen leakage outside the fovea. Endpoint is visual acuity and reduction of subretinal edema as determined by optical coherence tomography. Regarding AMD drusen maculopathy has to show soft confluent drusen and hyperpigmented spots. Angiographically a choroidal neovascularization has to be ruled out. Both eyes of the patient must have symmetric patterns since one eye is treated and the other one observed. End point would be a visual acuity and reduction of drusen as determined by fundus photography. For geographic atrophy due to age-related macular degeneration both eyes of the patient should present symmetric areas of atrophy. Laser treatment takes place at the rim of the atrophy zone in one eye whereas the other eye is observed. Due to RPE proliferation induced by SRT the major endpoint for this entity will be the stop or reduction of geographic atrophy enlargement in the treated eye compared with the fellow eye. Visual acuity should be at least 0.1.

All patients will be followed at various times after treatment as derived from a strict inclusion and follow-up protocol. The study is approved by the institutional study board and ethical committee; patients safety is covered by a private insurance company.

ELIGIBILITY:
Inclusion Criteria:

* symmetric drusen maculopathy with soft drusen both eyes
* symmetric geographic atrophy both eyes
* diabetic macular edema single eye
* acute or chronic central serous chorioretinopathy

Exclusion Criteria:

* previous laser treatment
* previous intravitreal injections
* choroidal neovascularization
* visual acuity > 0.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | up to 2 years

SECONDARY OUTCOMES:
drusen reduction | up to 2 years
area of geographic atrophy | up to 2 years
reduction of retinal edema | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Framme, MD, Principal Investigator — University Eye Hospital Regensburg
Locations (1):
- University Eye Hospital Regensburg, Regensburg, Germany